CLINICAL TRIAL: NCT01729546
Title: Evaluating System Accuracy of Blood Glucose Monitoring Systems for Self-testing in Managing Diabetes Mellitus [Following EN ISO 15197:2003 - 7.3 System Accuracy Evaluation] Part 40 of Study IDT-2010
Brief Title: Evaluating System Accuracy of Blood Glucose Monitoring Systems for Self-testing in Managing Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: IDT-1212
Record Dates: First submitted 2012-11-14; First posted 2012-11-20 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes
Keywords: SMBG (self-monitoring of blood glucose); POCT; System Accuracy
MeSH Terms: conditions — Diabetes Mellitus

INTERVENTIONS:
Device: 7 Blood glucose monitoring systems

SUMMARY:
In this clinical trial an evaluation of a blood glucose monitoring system (BGStar) and several POCT (point-of-care testing) devices against two laboratory methods will be performed. This evaluation will be performed according to ISO (International Organization for Standardization) 15197 System Accuracy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* People with diabetes Typ 1 or Typ 2 and people without diabetes
* for BG adjustment people with diabetes Typ 1 or Typ 2
* informed consent

Exclusion Criteria:

* pregnancy or lactation period
* severe acute diseases
* severe chronic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Evaluation of System Accuracy according to ISO 15197

CONTACTS AND LOCATIONS:
Locations (1):
- Institut für Diabetes-Technologie Forschungs- und Entwicklungsgesellschaft mbH an der Universität Ulm, Ulm, Germany

REFERENCES:
- [Result] Freckmann G, Schmid C, Pleus S, Baumstark A, Link M, Stolberg E, Haug C, Sieber J. System accuracy evaluation of systems for point-of-care testing of blood glucose: a comparison of a patient-use system with six professional-use systems. Clin Chem Lab Med. 2014 Jul;52(7):1079-86. doi: 10.1515/cclm-2013-0976. PMID 24681433
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/24681433